CLINICAL TRIAL: NCT04212715
Title: Prostate SABR With Intra-Prostatic SABR Boost: A Phase II Study
Brief Title: Prostate SABR With Intra-Prostatic SABR Boost
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr. Yasir Alayed, Consultant and Assistant Professor, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-19-4346
Record Dates: First submitted 2019-12-26; First posted 2019-12-27 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): SABR 35Gy/5 to prostate, up to 50Gy/5 to MR nodule, and 25Gy/5 to pelvic nodes and SVs
  Interventions: Radiation: Pelvic SABR with intra-prostatic SABR

INTERVENTIONS:
Radiation: Pelvic SABR with intra-prostatic SABR — SABR 25Gy / 5 fractions to pelvis; 35Gy / 5 fractions to prostate; up to 50Gy / 5 fractions to MR nodule

SUMMARY:
Stereotactic Ablative Radiation (SABR/SBRT) will be prescribed to a dose of 35 Gy in 5 fractions, once weekly to prostate with a simultaneous intra-prostatic boost to the MR detected nodule up to 50Gy. The pelvic lymph nodes and seminal vesicles will also receive 25 Gy in 5 weekly fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* High-risk prostate cancer, defined as at least one of: T3, Gleason 8-10, OR PSA > 20 ng/mL
* Willing to give informed consent to participate in this clinical trial

Exclusion Criteria:

* Prior pelvic radiotherapy
* Contraindication to radical prostate radiotherapy e.g. connective tissue disease or inflammatory bowel disease
* Contraindication to prostate MRI
* No evidence of castrate resistance (defined as PSA < 3 ng/ml while testosterone is < 0.7nmol/l. Patients could have been on combined androgen blockade but are excluded if this was started due to PSA progression.
* Definitive extrapelvic nodal or distant metastatic disease on staging investigations.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity | 3 month after accrual is completed
  To document the rate of acute urinary and bowel toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Alayed, MD, Principal Investigator — King Saud Medical City
Locations (1):
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No